CLINICAL TRIAL: NCT03664648
Title: HEPLISAV-B Pregnancy Registry: An Observational Study on the Safety of HEPLISAV-B Exposure in Pregnant Women and Their Offspring
Brief Title: DV2-HBV-27: Observational Pregnancy Registry
Acronym: HBV-27
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dynavax Technologies Corporation (Industry)
Collaborators: PPD, Part of Thermo Fisher Scientific (Industry)
Responsible Party: Sponsor
Other Study IDs: DV2-HBV-27
Record Dates: First submitted 2018-07-18; First posted 2018-09-10 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Pregnant
Keywords: Pregnant; Conceived; HBV Vaccine; Hepatitis B; Hepatitis B vaccine; HBV; Hepatitis; Registry; Prevention; Female volunteers
MeSH Terms: conditions — Hepatitis B; Hepatitis | interventions — Heplisav-B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Pregnant Women Exposed to HEPLISAV-B: Adult women who received a dose of HEPLISAV-B within 28 days prior to conception or at any time during pregnancy.
  Interventions: Biological: HEPLISAV-B

INTERVENTIONS:
Biological: HEPLISAV-B — This study is strictly observational. Administration of HEPLISAV-B, the schedule of office visits and all treatment regimens will be determined by the treating health care provider in the context of routine clinical care.

SUMMARY:
Purpose of the study is to evaluate pregnancy outcomes among women who received a dose of HEPLISAV-B within 28 days prior to conception or at any time during pregnancy

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* HEPLISAV-B exposure within 28 days prior to conception or at any time during pregnancy

Exclusion Criteria:

* Less than 18 years of age
* HEPLISAV-B exposure greater than 28 days prior to conception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Study Population: Women 18 years of age or older exposed to HEPLISAV-B within 28 days of conception or at any time during pregnancy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-21 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Congenital Malformations in Live-Born Infants. | Live-born infants will be followed to 12 months of age
Rate of Still Births, Pre-Term, or Fetal Loss (Including Spontaneous Abortion) of any Gestational Age | Follow-up will end at the time of pregnancy outcome up to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Registry Office, Recruiting Nationwide, Wilmington, North Carolina, United States